CLINICAL TRIAL: NCT01120613
Title: Post Kidney Transplant Nocturnal Hypertension Prevalence and Management Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: primary investigator left institution; not enough patients
Sponsor: Northwell Health (Other)
Responsible Party: Rajiv Vij MD MPH, North Shore LIJ
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-015A
Record Dates: First submitted 2010-04-29; First posted 2010-05-11 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension
Keywords: Nocturnal Hypertension; Nondipping; Renal Transplant; Chronotherapy
MeSH Terms: conditions — Hypertension | interventions — Chronotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chronotherapy (Experimental): Patients identified with Nocturnal Hypertension, will have one of the blood pressure medications switched from daytime dosing to nighttime dosing
  Interventions: Drug: Chronotherapy

INTERVENTIONS:
Drug: Chronotherapy — Patients identified with nocturnal hypertension while treated with blood pressure medications will have one medication switched from daytime to night time dosing in the following preference:
  1. ACE or ARB
  2. Calcium Channel Blockers
  3. Alpha Blocker
  4. Beta Blocker
  If patient is on only one daytime BP medication, it will be switched to night time dosing. No dose adjustments will be made nor any new medications will be added. Only timing of BP medication will be changed.

SUMMARY:
Hypertension (HTN) affects up to 75% of kidney transplant recipients and is associated with premature death. Nocturnal HTN is a common complication of ongoing essential HTN or a secondary cause of HTN. Both the non dipping of systolic blood pressure (SBP) at night time and the reverse dipping is associated with increased target organ damage and adverse cardiovascular outcomes and possibly allograft survival. Treatment of Nocturnal HTN is critical. Chronotherapy has been shown to be effective in halting progression in patients with diabetic nephropathy and chronic kidney disease. There is not enough data on prevalence and management of nocturnal HTN in transplant patients, which is the object of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant more than 1 year ago and not on dialysis.
2. Age between 18 years to 70 years.
3. Known history of HTN on one or more anti-hypertensive medication.
4. Stable anti-hypertensive regimen for past 2 months
5. One of the anti-hypertensive regimen must include an ACE inhibitor, or an angiotensin receptor blocker, calcium channel blocker, alpha or beta blocker.
6. Stable immunosuppressive regimen with no dose changes in past 3 months.
7. No hospitalizations for previous 2 months

Exclusion Criteria:

1. Inability to consent
2. History of falls
3. Presence of AVF or AVG in both the arms
4. Inability to follow up in renal transplant clinic.
5. History of Atrial fibrillation.
6. Pregnant Women
7. Parkinson's Disease
8. Severe orthostatic Hypotension
9. Severe autonomic dysfunction
10. History of other transplanted organs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Percent drop in mean SBP at night time compared to mean SBP at day time | 2 months

SECONDARY OUTCOMES:
Urine Microalbumin to creatinine ratio | 2 months
Change in Glomerular filtration rate as measured by MDRD equation. | 2 months
  Serum creatinine as a measure of kidney function will be measured at the begining and end of intervention.
24 hour mean systolic Blood Pressure (SBP) Control | 2 months
  Ambulatory Blood pressure monitoring at the end of intervention will be used to assess 24 hour ( day and nighttime) blood pressure control We hypothesize that night time dosing of medication ( chronotherapy) will not only improve nocturnal hypertension but also improve awake blood pressure and overall 24 hour average SBP control.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Vij, MD MPH, Principal Investigator — North Shore Long Island Jewish Hospital; Kenar Jhaveri, MD, Principal Investigator — North Shore Long Island Jewish Hospital
Locations (1):
- North Shore Long Island Jewish Hospital, Great Neck, New York, United States

REFERENCES:
- [Background] Paoletti E, Gherzi M, Amidone M, Massarino F, Cannella G. Association of arterial hypertension with renal target organ damage in kidney transplant recipients: the predictive role of ambulatory blood pressure monitoring. Transplantation. 2009 Jun 27;87(12):1864-9. doi: 10.1097/TP.0b013e3181a76775. PMID 19543066
- [Background] Paoletti E, Bellino D, Amidone M, Rolla D, Cannella G. Relationship between arterial hypertension and renal damage in chronic kidney disease: insights from ABPM. J Nephrol. 2006 Nov-Dec;19(6):778-82. PMID 17173252
- [Background] McGlothan KR, Wyatt RJ, Ault BH, Hastings MC, Rogers T, DiSessa T, Jones DP. Predominance of nocturnal hypertension in pediatric renal allograft recipients. Pediatr Transplant. 2006 Aug;10(5):558-64. doi: 10.1111/j.1399-3046.2006.00521.x. PMID 16856991
- [Background] Stenehjem AE, Gudmundsdottir H, Os I. Office blood pressure measurements overestimate blood pressure control in renal transplant patients. Blood Press Monit. 2006 Jun;11(3):125-33. doi: 10.1097/01.mbp.0000209080.24870.2d. PMID 16702821
- [Background] Oliveras A, Vazquez S, Hurtado S, Vila J, Puig JM, Lloveras J. Ambulatory blood pressure monitoring in renal transplant patients: modifiable parameters after active antihypertensive treatment. Transplant Proc. 2004 Jun;36(5):1352-4. doi: 10.1016/j.transproceed.2004.04.085. PMID 15251330
- [Background] Covic A, Segall L, Goldsmith DJ. Ambulatory blood pressure monitoring in renal transplantation: should ABPM be routinely performed in renal transplant patients? Transplantation. 2003 Dec 15;76(11):1640-2. doi: 10.1097/01.TP.0000091288.19441.E2. PMID 14702541
- [Background] Toprak A, Koc M, Tezcan H, Ozener IC, Oktay A, Akoglu E. Night-time blood pressure load is associated with higher left ventricular mass index in renal transplant recipients. J Hum Hypertens. 2003 Apr;17(4):239-44. doi: 10.1038/sj.jhh.1001536. PMID 12692568
- [Background] Hermida RC, Ayala DE. Chronotherapy with the angiotensin-converting enzyme inhibitor ramipril in essential hypertension: improved blood pressure control with bedtime dosing. Hypertension. 2009 Jul;54(1):40-6. doi: 10.1161/HYPERTENSIONAHA.109.130203. Epub 2009 May 11. PMID 19433778
- [Background] Hermida RC, Ayala DE, Fernandez JR, Calvo C. Chronotherapy improves blood pressure control and reverts the nondipper pattern in patients with resistant hypertension. Hypertension. 2008 Jan;51(1):69-76. doi: 10.1161/HYPERTENSIONAHA.107.096933. Epub 2007 Oct 29. PMID 17968001
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Chronotherapy with nifedipine GITS in hypertensive patients: improved efficacy and safety with bedtime dosing. Am J Hypertens. 2008 Aug;21(8):948-54. doi: 10.1038/ajh.2008.216. Epub 2008 Jul 3. PMID 18600215
- [Background] Hermida RC, Calvo C, Ayala DE, Lopez JE, Rodriguez M, Chayan L, Mojon A, Fontao MJ, Fernandez JR. Dose- and administration time-dependent effects of nifedipine gits on ambulatory blood pressure in hypertensive subjects. Chronobiol Int. 2007;24(3):471-93. doi: 10.1080/07420520701420683. PMID 17612946
- [Background] Minutolo R, Gabbai FB, Borrelli S, Scigliano R, Trucillo P, Baldanza D, Laurino S, Mascia S, Conte G, De Nicola L. Changing the timing of antihypertensive therapy to reduce nocturnal blood pressure in CKD: an 8-week uncontrolled trial. Am J Kidney Dis. 2007 Dec;50(6):908-17. doi: 10.1053/j.ajkd.2007.07.020. PMID 18037091
- [Background] Vij R, Peixoto AJ. Management of nocturnal hypertension. Expert Rev Cardiovasc Ther. 2009 Jun;7(6):607-18. doi: 10.1586/erc.09.42. PMID 19505276